CLINICAL TRIAL: NCT05759507
Title: Evaluation of Practices at the University Hospital of Nancy in the Context of Surgery During Pregnancy :a Retrospective Study Between 2014 and 2021
Brief Title: Evaluation of Practices at the University Hospital of Nancy in the Context of Surgery During Pregnancy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, TOURNIER Mathilde, Clinical director, Central Hospital, Nancy, France
Other Study IDs: 6030/2107
Record Dates: First submitted 2023-02-10; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Surgery; Pregnancy Complications; Pregnancy Related
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Women undergo pregnancy from 5 SA to 41 SA with no limitation of age
  Interventions: Procedure: abdominal surgery

INTERVENTIONS:
Procedure: abdominal surgery

SUMMARY:
About 2% of pregnant women are going through from surgery during pregnancy. These are mainly represented by emergencies like abdominal conditions such as appendicitis.

Pregnancy raises the issue of possible diagnostic confusion associated with operational difficulties related to a gravid uterus, i.e. increased in volume, and possible induced obstetric complications like premature delivery or miscarriage. late.

The management of these patients is therefore complex and the literature is poor on the subject.

DETAILED DESCRIPTION:
In the CHRU of Nancy because of the lack of guidelines, there is no guidelines on the management around urgent surgery during pregnancy.

The aim is to describe how patients on the 7 last years where taking care of and to examine if there where mistakes and delay due to pregnancy.'

The aim is also to describe the consequences of the surgery and analyse the end of the pregancy

ELIGIBILITY:
Inclusion Criteria:

* Women going through pregnancy

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women going through pregnancy with no limitation of age
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with no mistakes from the diagnosis to the surgery. | 1 year
  days of delay in the diagnosis ? error ? Diagnostic of certitude is established during surgery

SECONDARY OUTCOMES:
Impact on pregnancy | 1 year
  The impact on pregnancy is defined as the issues after surgery such as miscarries, premature labor, neonatal asphyxie etc..

CONTACTS AND LOCATIONS:
Locations (1):
- Maternite Regionale et Universitaire de Nancy, Nancy, Meurthe-et-moselle, France